CLINICAL TRIAL: NCT03444493
Title: The Effect of Stabilization Exercises on Pain, Disability and Physical Performance After Radiofrequency Lumbar Facet Denervation
Brief Title: The Effect of Stabilization Exercises After Radiofrequency Lumbar Facet Denervation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Research Assistant, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO14605
Record Dates: First submitted 2018-02-17; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Low Back Pain; Facet Joint Pain; Radiofrequency Denervation; Pain; Disability Physical
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Stabilizastion (exercise group) and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The exercise group performed specific localized exercises aimed at restoring the stabilizing protective function of the transversus abdominis (TrA). The exercises were designed specifically to activate and train the isometric holding function of the TrA muscle at the affected vertebral segment. Additionally, the exercise group was informed about protecting for biomechanics of lumbar spine.
  Interventions: Other: Exercise
- Control (No Intervention): Control group was informed about protecting for biomechanics of lumbar spine.

INTERVENTIONS:
Other: Exercise — Exercises were basically performed in 3 phases in this study. In the first phase; effectively and correctly contraction of TrA and multifidus muscles and how the patients adapted to daily life activities was taught. In the second phase; was aimed that the protection of stabilization by counteracting more muscle activation, in the third phase neutral position along with the activities required high level control.
  Arms: Exercise

SUMMARY:
A gap of knowledge exists on the understanding of the acute effects of stabilization exercises on pain, disability and physical performance when applied after radiofrequency denervation. Therefore, the main objective of this study is to show the effects of stabilization exercises when started in acute period and also reduce the frequency of recurrence low back pain of patients with FJS after radiofrequency denervation.

DETAILED DESCRIPTION:
Lumbar facet joint syndrome has been described as a potential cause of low back pain and affects an estimated 4% to 8% of those low back pain patients without neurological deficits or radiographic evidence of lumbar spine disease. The levels of physical performance and functional disability of the patients with lumbar FJS are affected because of the chronicity of the pain.

Radiofrequency denervation (RFD) is one of the therapautic procedures are used most commonly in treatment of facet joint syndrome. Numerous placebo-controlled trials have examined lumbar facet pain and demonstrated that RFD yields positive results in lumbar pain in properly selected patients. The lumbar stabilization exercise is based on the control of the local muscle system (multifidus, transversus abdominis, diaphragm and pelvic floor muscles) responsible for ensuring segmental stability of the vertebral colon in recent years.

In the clinical trials, stabilization exercises have been shown to reduce pain, improves physical performance and prevent the recurrent low back pain by strengthing of muscles supporting the vertebral colon.

Therefore, the main objective of this study is to show the effects of stabilization exercises when started in acute period and also reduce the frequency of recurrence low back pain of patients with FJS after radiofrequency denervation.

ELIGIBILITY:
Inclusion Criteria:

* age older than 45 year, failure to improve with conservative treatment, limited functions and daily life, pain exacerbated by rest, sitting or standing

Exclusion Criteria:

* previous surgical intervention in the spine or hip, previous local injection to the lumbar spine facet joint, current treatment with a narcotic drug, impairment of cognition or speech

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Change from Baseline visual analog scale(rest) after radiofrequency denervation (at 2 week) and after exercise procedure (at 8 week)
  Patients were asked to marked the level of pain on a 10 cm at rest, activity and sleep; VAS scale marked at one end as "no pain" and at the other as "worst pain imaginable''.
Visual Analog Scale | Change from Baseline visual analog scale(activity) after radiofrequency denervation (at 2 week) and after exercise procedure (at 8 week)
  Patients were asked to marked the level of pain on a 10 cm at activity; VAS scale marked at one end as "no pain" and at the other as "worst pain imaginable''.
Visual Analog Scale | Change from Baseline visual analog scale (sleep)after radiofrequency denervation (at 2 week) and after exercise procedure (at 8 week)
  Patients were asked to marked the level of pain on a 10 cm at sleep; VAS scale marked at one end as "no pain" and at the other as "worst pain imaginable''.

SECONDARY OUTCOMES:
Oswestry Disability Index | Change from Baseline Oswestry Disability Index after radiofrequency denervation (at 2 week) and after exercise procedure (at 8 week)
  The ODI assesses ten different aspects of disability (pain, personal care, lifting, sitting, standing, sleeping, sex life, social life, walking and travelling). Each parameter is scored from 0 to 5, with 0 indicating no functional limitation due to pain and 5 indicating a major functional disability due to low back pain. This questionnaire is scored using a global percentage score. The obtainable maximum score is 50, which corresponds to 100%.
Physical Performance | Change from Baseline physical performance tests after radiofrequency denervation (at 2 week) and after exercise procedure (at 8 week)
  Eight physical performance tests (PPT) of daily activities such as climbing stairs, picking up something from the floor, bending forward, rolling up from supine position, putting on a sock, standing up from a lying position etc. were evaluated. The tests were observed by trained physiotherapist, who judged the patients' individual performance in each test using four grades of movement quality that were recorded on a four-point ordinal scale (0; performs activity without any difficulty, 3; restricted movement: cannot perform activity).
Walking speed | Change from Baseline 10 meter walking speed after radiofrequency denervation (at 2 week) and after exercise procedure (at 8 week)
  10 meter walking speed was also measured and recorded as m/sec.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCormick ZL, Marshall B, Walker J, McCarthy R, Walega DR. Long-Term Function, Pain and Medication Use Outcomes of Radiofrequency Ablation for Lumbar Facet Syndrome. Int J Anesth Anesth. 2015;2(2):028. doi: 10.23937/2377-4630/2/2/1028. PMID 26005713
- [Background] Standaert CJ, Weinstein SM, Rumpeltes J. Evidence-informed management of chronic low back pain with lumbar stabilization exercises. Spine J. 2008 Jan-Feb;8(1):114-20. doi: 10.1016/j.spinee.2007.10.015. PMID 18164459